CLINICAL TRIAL: NCT00261807
Title: Open Label, Single Center Study to Evaluate Higher Doses of Daptomycin in the Treatment of Patients With Severe Necrotizing Skin and Soft Tissue Infections.
Brief Title: Daptomycin for the Treatment of Severe Necrotizing Soft-Tissue Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Denise Rudell, Program Manager for Dr. Manjari Joshi, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-26386
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Fasciitis, Necrotizing; Severe Necrotizing Skin and Soft Tissue Infections; Fournier's Gangrene
Keywords: severe; skin; infections
MeSH Terms: conditions — Fasciitis, Necrotizing; Soft Tissue Infections; Fournier Gangrene; Lymphoma, Follicular; Infections | interventions — Daptomycin

ARMS (1):
- Single ARM Study (Other): It was a single arm study with higher dose of daptomycin used for patients with severe skin and soft tissue infections.
  Interventions: Drug: Daptomycin 6mg/kg/day

INTERVENTIONS:
Drug: Daptomycin 6mg/kg/day

SUMMARY:
Daptomycin is a new antimicrobial agent which has activity against resistant Gram positive cocci including MRSA. The phase 3 clinical trials for skin and soft tissue infections (SSTI) with Staphylococci and Streptococci have already demonstrated that daptomycin was noninferior to the comparator agent (vancomycin or beta-lactams) (10). Although this clinical trial did not include any patients with clostridial infection, there is in vitro data to support the activity of daptomycin against a variety of clostridial species(11) ( Clostridium perfringens) Therefore, for this trial we will include patients with clostridial infections with this species. Additionally, the patients in the SSTI study were not as ill as the proposed study population. Therefore for treatment of such severe infections, we would like to use a higher dose of daptomycin (6mg/kg/dose). The reasons for using a higher dose of daptomycin in this subgroup are as follows:

1. Patients who are severely ill have an increased volume of distribution; and therefore have a lower serum concentration of daptomycin. These patients might require a higher dose of daptomycin to achieve the desired serum concentration.
2. One of the organisms involved in necrotizing fasciitis is enterococcus (both-fecalis and faecium). E.faecium has higher MICs to daptomycin and would require a higher dose of the drug to achieve adequate free (unbound) serum concentration of the drug.
3. Both necrotizing fasciitis and endocarditis are serious deep seated infections. The clinical trials for endocarditis are using 6mg/kg/dose of daptomycin.

Therefore for optimal treatment of necrotizing fasciitis, it is justifiable that we should use the higher dose of daptomycin.

Objective:

To evaluate the clinical and microbiological efficacy and safety of higher dose daptomycin therapy in the treatment of patients with severe necrotizing skin and soft tissue infections.

Type of Study:

Open label, single center study.

DETAILED DESCRIPTION:
At the shock trauma center, the management of patients with NSTI is conducted in the following fashion: All new patients with NSTI are admitted to the trauma center through the 12-bed shock trauma admitting area. Full hemodynamic resuscitation is undertaken. The on-call soft-tissue and infection team is mobilized. Standard investigations, radiographic evaluations, and laboratory tests, including gram stain and culture specimens, are obtained. The University of Maryland Medical Systems/shock trauma laboratory is utilized for hematology, biochemical, and bacteriologic studies. Aggressive empiric broad-spectrum antibiotic therapy is instituted. The standard antibiotic therapy for NSTI's at shock trauma includes the following:

Gram negative rods: Piperacillin/Tazobactam or quinolones or aztreonam /

+ aminoglycosides Anaerobes: Piperacillin/Tazobactam or Metronidazole or Clindamycin Gram positive cocci (not MRSA/VRE): Piperacillin/Tazobactam or Clindamycin Gram positive cocci (MRSA): Vancomycin Gram positive cocci (VRE): Linezolid For purposes of this study, daptomycin would replace Vancomycin, Linezolid or clindamycin for gram positive coverage. Prior antibiotic therapy, culture data, comorbid conditions, allergy history and other variables may result in institution of a different antibiotic regimen.

The patient is taken to the shock trauma operating room for debulking of infected tissue (excision and debridement) and reculturing. Postoperatively, the patient is moved to a critical or intensive care unit for further management and monitoring. When the patient is stable, HBO is begun within 12 hours of arrival. Once the patient is enrolled in the study the following procedures will be followed:

Antibiotic Therapy:

Once the patient is consented, the antibiotic therapy will be started. The combination regimen will include the following drugs in standard approved dosing.

* Gram negative bacteria: Aztreonam or ciprofloxacin / + aminoglycosides*
* Anaerobic bacteria: Metronidzole
* Gram positive bacteria: Daptomycin For all patients the recommended dose of Daptomycin will be 6 mgm/kg/day administered over 30 minutes. A pharmacokinetic study performed in obese patients demonstrated that daptomycin could be dosed based on total body weight. No adjustment in daptomycin dose should be required based solely on obesity (12). Any patient who develops a decrease in renal function during the study to the point where his/her creatinine clearance (CrCl) falls below 30 mL/min would have their dose adjusted to 6 mg/kg every 48 hours, the interval recommended by the package insert. This includes patients who go on to require conventional hemodialysis. Since there are no data available on the pharmacokinetics (PK) of daptomycin in patients receiving continuous renal replacement therapy (CRRT), and therefore no recommendation for dosage adjustment, these patients would be removed from the study and initiated on a standard of care regimen . Treatment duration will be 7-14 days.

  * Aminoglycosides will be added if there is suspicion or documentation of resistant gram negative rods.

At various intervals, the following information will be collected or procedures will be followed: (See attached study schedule) Baseline

1. Demographic data - age, gender, weight, height, nursing home residence
2. Number and length of previous hospitalizations in last six months
3. Nature and duration of symptoms
4. Admission status including vital signs, GCS, APACHE, SIRS scores, CBC with diff, CPK, lactate, BUN, creatinine, liver function tests, blood gases if on ventilator, cultures of wound-aerobic and anaerobic.
5. Prior surgery for NSTI - number and dates
6. Comorbid conditions - diabetes, peripheral vascular disease, immunocompromised, etc.
7. Prior antibiotics over last six months - dose/route/type
8. Prior cultures of NSTI, presence of resistant bacteria.
9. Wound size - length, depth in cm.
10. Use of drugs such as HMG-CoA reductase inhibitors

At various intervals, the following procedures will be followed:.

* GCS, vital signs, CBC, CPK, BUN, creatinine, liver functions, blood gases if ventilated
* Wound size in cm
* Surgical intervention
* Cultures of wound, (both aerobic and anaerobic), blood, super infections. Preferably cultures of the debrided tissue or purulent material will be obtained. If there is no tissue or pus available, only then a deep culture of the wound will be obtained. The culture will be evaluated in the microbiologic lab for gram stain, culture (aerobic and anaerobic if already indicated) and antimicrobiological sensitivity (by standard CLSI (NCCLS) techniques. The organisms in the study will be identified at the genus and species level.
* LOS - hospital, ICU
* Wound dressing - type
* Use of vacuum assisted dressing
* Duration of antibiotic therapy
* Adverse events
* Mortality
* Patient will be evaluated clinically on a daily basis by several clinical services (surgery, infectious diseases, critical care, hyperbaric medicine)and safety labs will be obtained every 3-5days. If a patient is failing therapy then based on available microbiological determinants, patient will be changed to an appropriate antibiotic regimen.

The End points of the study are as follows:

* clinical cure at 7-14 days
* clinical failure at any point after 72 hours of treatment
* if the patient is clinically cured and there is persistence of initial infective organism in the wound culture, the study would be terminated. However, if the patient is worse then appropriate treatment will be initiated and study drug will be discontinued.
* if the patient experiences a serious adverse event related to the study drug, the study drug will be terminated.
* if the patient decides to withdraw consent.

Clinical Response at the end of treatment (7-14 days) and test of cure (3-28 days) post end of treatment):

* Cure: Resolution of clinically significant signs and symptoms* associated with the infected wound present at the time of study entry and no additional gram-positive antibiotic therapy is needed until the end of treatment visit.
* Improved: Partial resolution of clinical signs and symptoms* of the wound (e.g., although the patient's clinical status has not completely returned to pre-infection baseline, the infectious process has been controlled) and no additional gram-positive antibiotic therapy is needed until the end of treatment visit.
* Failure: No response or worsening of clinical signs and symptoms of infection; or new signs and symptoms of infection are present; or additional gram-positive antibiotic therapy is needed until the end of treatment visit.
* Unable to Evaluate: Unable to determine response; e.g., no evaluation performed at the time point, or administration of non-study antibiotics effective against a study pathogen.

  * Clinically significant signs and symptoms are:
* pain out of proportion to clinical findings
* tenderness to palpation
* elevated temps.[100.4] or reduced temps.[>96]
* WBC counts > 12.000/cu.mm
* swelling
* erythema
* induration
* pus formation

Microbiological Response at End of Treatment and Test of Cure Visit:

* Documented Eradicated: The baseline infecting pathogen was absent at end of treatment as determined by a negative culture result.
* Presumed Eradicated: The baseline infection was presumed absent at the end of treatment as determined that there was "nothing to culture".
* Documented Persistent: The baseline infecting pathogen was present at the end of treatment.

Patients will also be monitored for 3 - 28 days post therapy.

Analysis Because of the small sample size (25 patients) stated above, this study will serve as a preliminary study to obtain data to evaluate the presence of positive trends in terms of outcome in the patients treated with Daptomycin. If favorable, this would warrant a larger prospective controlled study in which a larger sample size would allow for a more robust statistical analysis. Variables in the initial analysis will include antibiotic days, intensive care unit and hospital length of stay and mortality.

ELIGIBILITY:
Inclusion/Exclusion Criteria

Inclusion criteria :

1. Read and sign the consent form. If patient is unable to sign, the consent will be obtained from a legally authorized representative.
2. Male or female > 18 years of age
3. If female of child bearing potential, negative pregnancy test
4. Surgical diagnosis of severe necrotizing fasciitis, severe necrotizing skin and soft tissue infections (e.g. Fournier's gangrene)
5. A) At least three of the following clinical signs and symptoms of local infection should be present:

   * pain out of proportion to clinical findings
   * tenderness to palpation
   * swelling
   * erythema
   * induration
   * pus formation

   B) At least 1 of the two systemic conditions should be present:
   * Elevated temps.[100.4] or reduced temps. [<96]
   * WBC counts > 12.00/cu.mm
6. Positive gram stain or wound culture obtained within 3 calendar days prior to the first dose of Daptomycin.

   * positive gram stain would include gram positive cocci or gram positive rods
   * positive wound culture would include growth of staphylococci and/or streptococci and/or enterococcus and/or clostridia (Clostridium perfringens ).
7. If the patient is on HMG-CoA reductase inhibitors then these agents will be discontinued at the study initiation and resumed after discontinuation of daptomycin.

Exclusion criteria:

1. If female, pregnant, or lactating and breast-feeding
2. Previous antibiotic therapy exceeding 72 hours duration, unless patient is worsening clinically or has gram positive pathogens cultured from wound that are resistant to current antibiotic therapy.
3. Sites of infection other than skin i.e., osteomyelitis, meningitis, bacteremia, etc.
4. Known to be allergic or intolerant to study medications
5. Expected to die in < 5 days
6. Significant renal impairment - creatinine clearance < 30m/min
7. A primary diagnosis of uncomplicated skin infections, such as cellulitis, minor post-op. wound infection, small decubitus ulcer etc.
8. Patients with baseline CPKs equal to or greater than 10 times upper limit of normal without myopathy and CPK elevation of greater than or equal to 5 times upper limit of normal with symptoms of myopathy
9. Documentation of myoglobinuria at onset of the study. The study will be conducted over a one-year period. We are anticipating enrollment of 25 patients on the study.

Criteria for withdrawal from the study:

1. If the patient complains of myalgias and has high CPK values as specified below.
2. If the patient develops myoglobinuria, CPKs equal to or 10 times upper limit of normal without myopathy and CPK elevation of greater than 5 times upper limit of normal with symptoms of myopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manjari G Joshi, MD, Principal Investigator — University of Maryland, School of Medicine - Shock Trauma
Locations (1):
- R Adams Cowley Shock Trauma Center, U. of Maryland Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from an academic inpatient center which sees about 200 severe soft tissue patients every year. Subjects were enrolled from (2005-2008).
Pre-assignment Details: Patients with necrotizing skin infections were screened for the study. A total of 25 subjects were enrolled. Patients were excluded if they had renal failure, high CPK, or myoglobln or if they did not meet the inclusion exculsion criteria. Also, if patient was unable to give consent and family was not present.
Groups:
- Single ARM Study: It was a single arm study with daptomycin use at a higher dose for patients with severe skin and soft tissue infections.
  Daptomycin 6mg/kg/day
Period: Overall Study
Arm/Group | Single ARM Study
Started | 25
Completed | 18
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Patients with severe necrotrotizing skin infections requiring surgical debridement, as well as antimicrobial therapy.
Arm/Group | Single ARM Study
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — No additional information.
  participants
    United States | 25
WBC Counts,Fever and Wound Appearance. [Number; unit: participants] — WBC counts of > 12 (cu/mm) were recorded. Fever was recorded: more than 100.4F or reduced temps < 96F
  Wound erythema, induration/swelling, and suppuration were visually noted as absent or present.
  Please note these are mostly subjective clinical findings of a wound exam.
  participants | 25

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to High Dose Daptomycin Therapy at End of Treatment (EOT)
Description: Clinical response was assessed by measuring impact of therapy on certain wound parameters. Specifically Erythema, Induration/Swelling, Suppuration, were recorded visually and WBC Counts were considered improved if <12,000/cu mm.
  The clinical response was documented as:
  1. CURE (resolution of clinical signs and symptoms and no additional need for gram-positive antibiotic therapy.
  2. IMPROVED (partial resolution of clinical signs and symptoms (although patient's clinical status had not completely returned to preinfection baseline but infectious process had been controlled , no additional gram-positive antibiotic therapy was needed;
  3. FAILURE (no response, worsening of clinical signs and symptoms of infection; or additional gram-positive antibiotic therapy was needed );
  4. UNABLE TO EVALUATE (unable to determine response; e.g., no evaluation performed at specified time points, or administration of non-study antibiotics effective against study pathogen).
Time Frame: The clinical response was measured at the end of treatment (7-14 days)
Population: Of the total 25 patients enrolled, 18 were measured as described in Baseline Population
Measure: Count of Participants; unit: Participants
Arm/Group | Single ARM Study
Number analyzed (Participants) | 18
Participants
  Erythema-EOT: Cure | 16
  Erythema-EOT: Improved | 0
  Erythema-EOT: Failure | 2
  Erythema-EOT: Unable to Evaluate | 0
  Induration EOT: Cure | 17
  Induration EOT: Improved | 0
  Induration EOT: Failure | 1
  Induration EOT: Unable to Evaluate | 0
  Suppuration-EOT: Cure | 13
  Suppuration-EOT: Improved | 0
  Suppuration-EOT: Failure | 5
  Suppuration-EOT: Unable to Evaluate | 0
  WBC Counts EOT: Cure | 18
  WBC Counts EOT: Improved | 0
  WBC Counts EOT: Failure | 0
  WBC Counts EOT: Unable to Evaluate | 0

2. Primary Outcome: Clinical Response to High Dose Daptomycin Therapy at Test of Cure (TOC)
Description: as for outcome 1
Time Frame: The clinical response was measured at Test of Cure (3-28 days post end of treatment)
Population: Of the total 25 patients enrolled, 18 were measured as described in Baseline Population
Measure: Count of Participants; unit: Participants
Groups:
- Single ARM Study: It was a single arm study with higher dose of daptomycin used for patients with severe skin and soft tissue infections.
  Daptomycin 6mg/kg/day
Arm/Group | Single ARM Study
Number analyzed (Participants) | 18
Participants
  Erythema-TOC: Cure | 18
  Erythema-TOC: Improved | 0
  Erythema-TOC: Failure | 0
  Erythema-TOC: Unable to Evaluate | 0
  Induration TOC: Cure | 18
  Induration TOC: Improved | 0
  Induration TOC: Failure | 0
  Induration TOC: Unable to Evaluate | 0
  Suppuration: Cure | 18
  Suppuration: Improved | 0
  Suppuration: Failure | 0
  Suppuration: Unable to Evaluate | 0
  WBC Counts-TOC: Cure | 18
  WBC Counts-TOC: Improved | 0
  WBC Counts-TOC: Failure | 0
  WBC Counts-TOC: Unable to Evaluate | 0

3. Secondary Outcome: Microbiological Response to High Dose Daptomycin Therapy at End of Treatment (EOT) and Test of Cure (TOC)
Description: Bacterial cultures were obtained in all patients and repeated if the patient had a second surgical intervention.
  The microbiological responses were documented as follows:
  1. DOCUMENTED ERADICATED: the baseline infecting pathogen was absent at end of treatment as determined by a negative culture.
  2. PRESUMED ERADICATED: The baseline infection was presumed absent at the end of treatment as determined that there was "nothing to culture".
  3. DOCUMENTED PERSISTENT: The baseline infecting pathogen was present at the end of treatment.
Time Frame: The microbiologicall response will be measured at the end of treatment (7-14 days) and Test of Cure (TOC) (3-28 days)
Population: Of the 25 patients enrolled in study, 23 were analyzed for Microbiological response at end of treatment and only 18 analyzed at Test of Cure visit (2 lost to follow up, 2 received additional antibiotics for infections at other sites (unrelated to primary infection) and 1 patient died during the study period)
Measure: Count of Participants; unit: Participants
Arm/Group | Single ARM Study
Number analyzed (Participants) | 23
Participants
  End of Therapy: Documented Eradicated | 0
  End of Therapy: Presumed Eradicated | 23
  End of Therapy: Documented Persistent | 0
  Test of Cure: number analyzed (Participants) | 18
  Test of Cure: Documented Eradicated | 0
  Test of Cure: Presumed Eradicated | 18
  Test of Cure: Documented Persistent | 0

ADVERSE EVENTS:
Time Frame: From initiation of study until Test of Cure (defined as 3-28 days from end of treatment, which was an average duration of 9.4 days of therapy, with a range between 7 and 14 days)
Description: Events described consistent with clinicaltrials.gov definitions
Arm/Group | Single ARM Study
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single ARM Study (N=25)
Gram Negative Rod Bacteremia (Infections and infestations) | 1 (1) — One patiient developed central line related bacteremia with acinetobacter.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single ARM Study (N=25)
C. difficle infection (Infections and infestations) | 1 (1) — C. difficle diarrhea
Vaginal Yeast Infection (Infections and infestations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3) — Anemia
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash
Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Swelling of lower extremity
High CPK (General disorders) | 1 (1) — High CPK Level

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No